CLINICAL TRIAL: NCT05119699
Title: An Open-label Trial on Accelerated Sequential Bilateral Theta Burst Repetitive Transcranial Magnetic Stimulation in Treatment-resistant Late-life Depression
Brief Title: Accelerated TBS in Late Life Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070-2021
Record Dates: First submitted 2021-10-22; First posted 2021-11-15 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Treatment Resistant Depression
Keywords: Treatment Resistant Depression; rTMS; Accelerated TBS; Late Life Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: This study is a single-arm, open-label, feasibility trial for the assessment of the clinical effects of a course of accelerated bilateral sequential TBS for LLD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active rTMS treatment (Experimental): Patients will receive accelerated TBS
  Interventions: Device: MagPro X100/R30 stimulator equipped with the B70 fluid-cooled coil

INTERVENTIONS:
Device: MagPro X100/R30 stimulator equipped with the B70 fluid-cooled coil — Subjects will receive 5 consecutive days (always Monday to Friday) of TBS rTMS, administered 8 times daily at 1 hour intervals. Patients will undergo cTBS of the R DLPFC at 110-120% RMT using bursts of 3 pulses at 50 Hz, bursts repeated at 5 Hz for a total of 600 pulses over 40 seconds, followed by iTBS of the L DLPFC at 110-120% resting motor threshold (RMT) using bursts of 3 pulses at 50 Hz, bursts repeated at 5 Hz with a duty cycle of 2 s on, 8 s off for a total of 600 pulses over 3 min 9 s. Participants will be titrated to 110-120% RMT within the first four treatments to aid with tolerability. If patients tolerate the stimulation well, the target will be 120%. Assessments focused on depressive symptoms will be administered at baseline, after final treatment and four weeks post final treatment.

SUMMARY:
This study is a single-arm, open-label, feasibility trial for the assessment of the clinical effects of a course of accelerated bilateral sequential theta burst stimulation (TBS) for late life depression (LLD). Over approximately 1 year, 30 outpatients at the Centre for Addiction and Mental Health (CAMH) meeting diagnostic criteria for LLD will be recruited and will receive 5 consecutive days (always Monday to Friday) of TBS repetitive transcranial magnetic stimulation (rTMS), administered 8 times daily at approximately 1 hour intervals, with continuous theta-burst stimulation (cTBS) applied to the right dorsolateral prefrontal cortex (DLPFC) followed by left DLPFC intermittent theta-burst stimulation (iTBS).

Patients will undergo a series of assessments as well as motor threshold testing to determine the appropriate site and strength of stimulation according to standard methods and then begin treatment.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an evidenced based treatment for medically refractory major depressive disorder (MDD). rTMS involves direct stimulation of cortical neurons using externally applied, powerful, focused magnetic field pulses. Dozens of studies and several meta-analyses over the last 15 years have shown that rTMS of the dorsolateral prefrontal cortex (DLPFC) produces statistically significant improvements in MDD, even when medications have failed. In the most recent generation of randomized controlled trials, rTMS consistently achieves response rates of 50-55% and remission rates of 30-35% in medically refractory MDD patients. rTMS has been shown to be effective and well tolerated for depression in younger and older adults. However, early rTMS studies with older adults were limited by suboptimal stimulation parameters, small sample sizes and insufficient treatment durations. The optimal parameters for rTMS are still in the process of being established, however the most widely-used rTMS protocols apply excitatory, 10 Hz stimulation to the left DLPFC; high frequency left (HFL) or inhibitory, 1 Hz stimulation to the right DLPFC; low frequency right (LFR), or both. Taken together with the reported findings of several other groups, results suggest that accelerated rTMS may be feasible, tolerable, and capable of achieving comparable and potentially better remission rates than longer 20 to 30 day courses. However, all of these studies were small, open-label case series, focused on younger adults.

ELIGIBILITY:
Inclusion Criteria:

1. Are voluntary and competent to consent to treatment
2. are an outpatient
3. are ≥60 years old
4. have a Mini-International Neuropsychiatric Interview (MINI 6.0) confirmed diagnosis of major depressive disorder (MDD), with a current major depressive episode (MDE)
5. have failed to achieve a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score of > 3 in the current episode or have failed to tolerate two separate trials of an antidepressant
6. have a score > 18 on the Montgomery-Asberg Depression Rating Scale (MADRS)
7. have had no increase or initiation of any antidepressant or antipsychotic medication in the 4 weeks prior to screening
8. Pass the TMS adult safety screening (TASS) questionnaire

Exclusion Criteria:

1. have a history of substance dependence or abuse within the last 3 months
2. have a concomitant major unstable medical illness as determined by one of the study physicians
3. have active suicidal intent
4. have a lifetime MINI diagnosis of bipolar I or II disorder, or primary psychotic disorder
5. have current psychotic symptoms
6. have a diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia, assessed by a study investigator to be primary. One of these comorbidities will not be exclusionary if they are not deemed to be primary.
7. have a diagnosis of any personality disorder as assessed by a study investigator to be primary and causing greater impairment than MDD
8. have presumed or probable dementia or clinical evidence of dementia as assessed by a Short Blessed Test score of greater than 10.
9. did not respond to a course of electroconvulsive therapy (ECT) in the current depressive episode
10. have received rTMS in the current episode, patients who have had rTMS in a previous episode would be eligible
11. have a history of a primary seizure disorder or a seizure associated with an intracranial lesion.
12. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
13. have a implanted electronic device that is currently function such as a defibrillator
14. currently take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant
15. if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
16. non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-10-14 (Estimated); Study Completion 2023-10-14 (Estimated)

PRIMARY OUTCOMES:
Changes in Montgomery-Asberg Depression Rating Scale (MADRS) score | baseline, last day of treatment (day 5, after the final treatment) and 4 weeks post treatment
  The investigators will assess the effects of accelerated sequential bilateral TBS based on change on the MADRS using an ANCOVA covarying for baseline differences to measure the change at the final time point for each subject. Higher MADRS scores indicates more severe depression. The overall score ranges from 0 to 60.

SECONDARY OUTCOMES:
Changes in 17 Item Hamilton Rating Scale for Depression (HDRS-17) | baseline, last day of treatment (day 5, after the final treatment) and 4 weeks post treatment
  The investigators will assess the effects of accelerated sequential bilateral TBS based on change on the HDRS-17 using an ANCOVA covarying for baseline differences to measure the change at the final time point for each subject. Higher HDRS-17 scores indicates more severe depression. The overall score ranges from 0 to 53.
Changes in Beck Depression Inventory (BDI-II) | baseline, last day of treatment (day 5, after the final treatment) and 4 weeks post treatment
  The investigators will assess the effects of accelerated sequential bilateral TBS based on change on the BDI-II using an ANCOVA covarying for baseline differences to measure the change at the final time point for each subject. Higher BDI-II scores indicates more severe depression. The overall score ranges from 0 to 63.
Changes in Beck Suicide Scale for Suicide Ideation (BSS) | baseline, last day of treatment (day 5, after the final treatment) and 4 weeks post treatment
  The investigators will assess the effects of accelerated sequential bilateral TBS based on change on the BSS using an ANCOVA covarying for baseline differences to measure the change at the final time point for each subject. Higher BSS scores indicates more severe suicidality. The overall score ranges from 0 to 38.
Changes in General Anxiety Disorder-7 (GAD-7) | baseline, last day of treatment (day 5, after the final treatment) and 4 weeks post treatment
  The investigators will assess the effects of accelerated sequential bilateral TBS based on change on the GAD-7 using an ANCOVA covarying for baseline differences to measure the change at the final time point for each subject. Higher GAD-7 scores indicates more severe anxiety. The overall score ranges from 0 to 21.

CONTACTS AND LOCATIONS:
Overall Officials: Alisson Trevizol, MD, Principal Investigator — CAMH
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hui J, Trevizol AP, Lee HH, Zomorrodi R, Zrenner C, Mulsant BH, Blumberger DM. Effects of Comorbid Anxiety on Treatment Outcomes After Accelerated Theta Burst Stimulation for Late-Life Depression. Am J Geriatr Psychiatry. 2026 Feb;34(2):229-234. doi: 10.1016/j.jagp.2025.09.017. Epub 2025 Sep 20. PMID 41109788